CLINICAL TRIAL: NCT01722760
Title: AD-ON: The Danish Study on Tidal Neonatal Nitrogen Oxide (NO) and Vitamins A and D as Possible Predictors of BPD
Brief Title: Tidal Neonatal NO, Vitamins A and D, and Infant Lung Disease - The AD-ON Study
Status: Completed | Type: Observational
Sponsor: Hillerod Hospital, Denmark (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Birgitte Johanne Schmidt, MD, Hillerod Hospital, Denmark
Other Study IDs: H-4-2012-091
Record Dates: First submitted 2012-10-24; First posted 2012-11-07 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Term Delivery With Preterm Labor, Third Trimester; Term Delivery With Preterm Labor, Unspecified Trimester; Bronchopulmonary Dysplasia
Keywords: Neonatal; Preterm; Bronchopulmonary Dysplasia; Nasal Continuous Positive airway Pressure (CPAP); Oxygen; Vitamin A; Vitamin D; Nitrogen oxide (NO); Reference material
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Air samples for Nitrogen oxide NO. Maternal, cord and neonatal blood samples for vitamins A and D.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Term and preterm infants: Term and preterm infants
  Interventions: Procedure: measurements

INTERVENTIONS:
Procedure: measurements

SUMMARY:
Children born prematurely are of greater risk of developing chronic lung disease (Bronchopulmonary Dysplasia).

With an increase in the amount of premature children, we expect an increasing number of children with BPD.

Today we do not have many ways of predicting or treating this condition, and the children are usually in hospital for several months after birth. Many are dismissed with home oxygen. Children with BPD are typically often re-submitted to hospital with respiratory disease the first couple of years, and some of them have problems throughout childhood and into adulthood.

Other scientists have found a correlation between BPD and Chronic Obstructive Pulmonary Disease (COPD).

The condition as well as the treatment (steroids), are associated with great risk of adverse effects as Cerebral Palsy, blindness, deafness and mental retardation.

The investigators wish to find a safe way to identify the children in greater risk of developing BPD, who could therefore benefit from a more intensive treatment.An early diagnosis would increase the possibility of predicting the prognosis.

Other studies have proven a connection between both low vitamin A and D and high exhaled nitrogen oxide (NO) with lung disease.

With this trial the investigators wish to make a reference material for NO and vitamins A and D in infants admitted to the neonatal department at two hospitals in Denmark, both with and without treatment with nasal Continuous Positive Airway Pressure.

The investigators furthermore wish to describe an eventual connection between BPD and these factors by examining a large group of children on 7 specific occasions within the first two months of life and at a one year follow up.

ELIGIBILITY:
Inclusion Criteria:

Cohort inclusion - All term and preterm infants admitted to Neonatal (Intensive) Care Unit. Gestational Age 24-42 weeks.

Exclusion Criteria:

1. Children with ciliary dyskinesia, as NO is distinguishable lower in these children.
2. Children who can not cooperate to the examination.
3. Children so dependant on oxygen, that the examination/measurement is not possible.
4. Children with pneumothorax
5. Children having a diagnosed pneumonia verified by tracheal secrete.
6. Children with bigger congenital anomalies

Max Age: 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term and preterm infants admitted to Neonatal Care Unit for reference material as control group.
  Preterm infants admitted to Neonatal Intensive Care Unit developing BPD as study group.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2013-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Tidal exhaled Nitrogen Oxide | 6-7 measures within the first 2 months of life and at 1 year of age.
  Reference material of tidal expiratory NO in a cohort of neonates admitted to Neonatal Intensive Care Unit and Neonatal Care Unit will be made.
  All children in the study will be measured on 8 occasions including a one year follow up.
  Association with Bronchopulmonary Dysplasia (BPD) and the measures above will be noted.

SECONDARY OUTCOMES:
Vitamin levels | From birth to a one year follow up
  Blood levels of Vitamins A (s-retinol) and D (se-25(OH)D2 and D3) will be measured at 3 preset occasions and at one year follow up, as well as maternal and cord blood at the time of birth.
  Reference material will be made and association to BPD will be noted.

OTHER OUTCOMES:
Bronchopulmonary Dysplasia | From premature birth to a one year follow up
  The incidence of BPD and the correlation the the above mentioned biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte J Schmidt, MD, Principal Investigator — Children´s Dep, North Zealand Hospital Hilleroed, Denmark
Locations (2):
- Denmark (2):
  - Neonatal departement GN, Rigshospitalet, Copenhagen, Region H
  - Children´s Departement, North Zealand Hospital, Hilleroed, Hilleroed, Region H